CLINICAL TRIAL: NCT04228523
Title: Therapeutic Education in Parkinson's Disease: What Impact on Drug Representations of Patients?
Brief Title: Therapeutic Education in Parkinson's Disease: What Impact on Drug Representations of Patients? (ETPARK-REMED)
Acronym: ETPARK-REMED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: France Parkinson Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/19/0183; 2019-A02754-53 (Other: ID-RCB)
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2023-08

CONDITIONS: Parkinson Disease
Keywords: Therapeutic education; Parkinson Disease; Socials representations
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: therapeutic education or speaking group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic education workshop (Experimental): Two group receive therapeutic education workshop already existing in Toulouse University Hospital
  Interventions: Other: Therapeutic education workshop
- Speaking Therapy (Other): One group receive speaking therapy already existing in Toulouse University Hospital
  Interventions: Other: Speaking Therapy

INTERVENTIONS:
Other: Therapeutic education workshop — Workshop on Parkinson disease drug has several educative sequences (lasting 4hours).
  * A first round table is organized to know the needs and issues related to drug management of patients.
  * The 1st educative sequence consists in knowing the different class of dopaminergic drugs and their action.
  * The 2nd educative sequence leads patients to understand their prescription and be aware of the needs to take pills regularly.
  * The 3rd educative sequence consists in learning and identifying potentials adverse effects and finds effective strategies to prevent them.
  At the end, one patient explains its tips and tricks about its drug management
  Arms: Therapeutic education workshop
Other: Speaking Therapy — Speaking group is leaded by a psychologist from Centre Expert Parkinson (lasting 2 hours). This specific time is an exchange between patients with Parkinson disease who feel free to come. It is about sharing its own experience. It is a very special moment, confidential and kindly where patients don't judge themselves and speak only if they want to.
  Arms: Speaking Therapy

SUMMARY:
Dopaminergic drug can have adverse effects leading to potential serious consequences. Therapeutic patient education must promote the understanding of drugs to improve its management. This study tries to evaluate the effect of therapeutic education workshop on Parkinson disease's drug (drug workshop) on the evolution of drug's representations in patients with Parkinson's disease compared to a control group.

DETAILED DESCRIPTION:
Dopaminergic drug can have adverse effects leading to potential serious consequences. Therapeutic patient education must promote the understanding of drugs to improve its management.

The therapeutic educational program ETPARK includes individual's consults or workshop. The team frequently offer to patients to participate in workshop on Parkinson disease's drug.

This study tries to evaluate the effect of therapeutic education workshop on Parkinson disease's drug (drug workshop) on the evolution of drug's representations in patients with Parkinson's disease compared to a control group (speaking group) at 1 and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's disease according to the United Kingdom Parkinson Disease Society Brain Bank (UKPDSBB) criteria,
* Patients who are already in therapeutic education program ETPARK,
* Patients who need and want to participate in therapeutic education workshop on Parkinson disease drug,
* Patients with health insurance,
* Patients who have signed a written informed consent form.

Exclusion Criteria:

* Patients suffering from another parkinsonian syndrome (multiple system atrophy, progressive supranuclear palsy etc.),
* Patients who has already done workshop on Parkinson disease drug (program ETPARK)
* Patients already included in clinical trial during the study,
* Patients who have severe psychiatric disorders or dopaminergic psychosis,
* Patients with cognitive impairment,
* Patients unable to complete the various scales used in the study,
* Patients under juridical protection,
* Women pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Evolution of Drug representation in Patients : BMQ | Three months
  Evolution of Drug representation through the Believe about Medicines Questionnaire (BMQ) compared to the control group. Evolution will be compared between the Baseline and the end of the study
  BMQ with eighteen items coded from 1 " "strongly agree" to 5 "strongly disagree".
Evolution of Drug representation in Patients : Verbal association | Three months
  Evolution of Drug representation through verbal association tasks compared to the control group. Evolution will be compared between the Baseline and the end of the study

SECONDARY OUTCOMES:
Drug representation in caregivers : Verbal association | Day 1
  Drug representation through verbal association tasks.
Drug representation in caregivers : BMQ | Day 1
  Drug representation through the Believe about Medicines Questionnaire (BMQ). BMQ with eighteen items coded from 1 " "strongly agree" to 5 "strongly disagree".
Knowledge about the disease | three months
  Evolution between Baseline and three months with a test created for the study. The test have 8 questions with two answers possible : True or False
Evolution in life quality : VAS | three months
  Evolution in life quality evaluate with Visual Analog Scale (VAS), 0 being the worst quality of life and 10 the best quality of life he can have.
  Evolution between Baseline and three months
Evolution in life quality : PDQ-(39) | three months
  Evolution in life quality evaluate with Parkinson Disease Quotation (PDQ)-39 with thirty-nine items coded from 1 " "always" to 5 "never". The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people affected by Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication.
  Evolution between Baseline and three months

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brefel-Courbon, MD, Principal Investigator — Univeristy Hospital Toulouse
Locations (1):
- Toulouse University Hospital, Toulouse, Occitanie, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canivet C, Costa N, Ory-Magne F, Arcari C, Mohara C, Pourcel L, Derumeaux H, Berard E, Bourrel R, Molinier L, Brefel-Courbon C. Clinical Impact and Cost-Effectiveness of an Education Program for PD Patients: A Randomized Controlled Trial. PLoS One. 2016 Sep 29;11(9):e0162646. doi: 10.1371/journal.pone.0162646. eCollection 2016. PMID 27685455
- [Background] Ory Magne F, Arcari C, Canivet C, Sarrail M, Fabre MH, Mohara C, Brefel Courbon C. [A therapeutic educational program in Parkinson's disease: ETPARK]. Rev Neurol (Paris). 2014 Feb;170(2):128-33. doi: 10.1016/j.neurol.2013.08.007. Epub 2013 Nov 20. French. PMID 24267951
- [Result] Faurie I, Harroch E, Scotto d'Apollonia C, Corte S, Arcari C, Mohara C, Barthelemy C, Fabre MH, Boussac M, Damase-Michel C, Almudever B, Croity-Belz S, Brefel-Courbon C. Impact of therapeutic education on the evolution of social representations of medication in patients with Parkinson's disease: A quantitative and qualitative study (ETPARK REMED). Rev Neurol (Paris). 2023 Dec;179(10):1086-1094. doi: 10.1016/j.neurol.2023.03.026. Epub 2023 Aug 24. PMID 37633737